CLINICAL TRIAL: NCT03588325
Title: Evaluation of MDW for Early Detection of Sepsis In the Emergency Department
Brief Title: Evaluation of MDW for Early Detection of Sepsis, Clinical Validity
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C26841
Record Dates: First submitted 2018-07-06; First posted 2018-07-17 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Severe Infection; Sepsis; Severe Sepsis
Keywords: MDW; Sepsis
MeSH Terms: conditions — Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples from LPS to be stored frozen for subsequent testing for sepsis biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CBC-DIFF with MDW, PCT, CRP — Tests will be run to determine early identification of sepsis and added value of the combination of tests. Results will not be used to manage patients

SUMMARY:
The purpose of this study is to confirm the clinical validity and the performance of the Monocyte Width Distribution (MDW) parameter to detect the development of sepsis in a prospective study of Emergency Department (ED) adults who have blood draw including Complete Blood Count with differential (CBC-DIFF) ordered upon presentation in a Spanish & French hospital and to verify cut-off for Tri-potassium ethylenediaminetetraacetic acid (K3EDTA).

DETAILED DESCRIPTION:
To confirm the clinical validity and performance of the Monocyte Width Distribution (MDW) parameter to detect the development of sepsis in a prospective study of ED adults who have blood draw including CBC with Differential ordered upon ED presentation. Septic patients are identified as those with values equal to or above the MDW threshold and non-septic patients are those with MDW values below the threshold. As the anticoagulant used at the sites is K3EDTA, the cut-off value will be assessed using sepsis cases and all corresponding non-sepsis to confirm optimal cut-off.

To explore the added value of this parameter in a patient diagnostic pathway that includes the use of procalcitonin (PCT) or C reactive protein (CRP) for the identification of septic patients All enrolled subjects will have PCT/ CRP assay performed per protocol Plasma will be aliquot and stored frozen for subsequent testing at Beckman Coulter for other sepsis biomarker tests (additional PCT& CRP tests and interleukin-6 (IL-6) on the sponsor's devices

ELIGIBILITY:
Inclusion Criteria:

* CBC-DIFF upon presentation
* Adults (18-89) of all races & ethnicities
* Signed Informed Consent

Exclusion Criteria:

* Previously enrolled
* Incomplete Informed Consent
* Subject discharged <4 hours from presentation
* PCT or CRP not performed per protocol
* Pregnancy
* Prisoners
* Subjects Under Custody or Guardianship

Ages: 18 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adults with suspicion of infection who present to the Emergency Department and for whom a CBC-DIFF is ordered upon presentation
Sampling Method: Probability Sample
Enrollment: 947 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Identification of sepsis based on Sepsis-2 criteria | Within 4 hours of presentation
  Determination of diagnostic accuracy based on Receiver Operating Characteristic Curves

SECONDARY OUTCOMES:
Identification of sepsis based on Sepsis-3 criteria | Within 4 hours of presentation
  Determination of diagnostic accuracy based on Receiver Operating Characteristic Curves

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Hausfater, MD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (2):
- La Pitié-Salpétrière, Paris, France
- Hospital Universitari Germans Trias I Pujol, Badalona, Spain

REFERENCES:
- [Derived] Hausfater P, Robert Boter N, Morales Indiano C, Cancella de Abreu M, Marin AM, Pernet J, Quesada D, Castro I, Careaga D, Arock M, Tejidor L, Velly L. Monocyte distribution width (MDW) performance as an early sepsis indicator in the emergency department: comparison with CRP and procalcitonin in a multicenter international European prospective study. Crit Care. 2021 Jun 30;25(1):227. doi: 10.1186/s13054-021-03622-5. PMID 34193208